CLINICAL TRIAL: NCT01829672
Title: Non-invasive Diagnostics of Pulmonary Hypertension With Dual Energy Computed Tomography - Prospective Study
Brief Title: Non-invasive Diagnostics of Pulmonary Hypertension With Dual Energy Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Ludwig Boltzmann Gesellschaft (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-174 ex 12/13
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Early diagnosis of pulmonary arterial hypertension; dynamic dual-energy computed tomography
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Other: pulmonary vascular disease (Experimental): Dual-energy computed tomography investigation
  Interventions: Radiation: Dual-energy computed tomography investigation

INTERVENTIONS:
Radiation: Dual-energy computed tomography investigation — 1x 20ml Ultravist (370mg J/ml)3-5ml/s, i.v.
  1x 40ml Ultravist (370mg J/ml)3-5ml/s i.v. Contrast agent administration
  Other Names: CT

SUMMARY:
The aim of the study is to determine relevant hemodynamic parameters for the diagnostics of pulmonary arterial hypertension (PAH) by dynamic contrast enhanced dual-energy CT (DE-CT). In this prospective study the investigators validate DE-CT results of patients against hemodynamic parameters from right heart catheterisation and control the results by other clinical investigations. The investigators expect that using this non-invasive method, parameters relevant for the diagnosis of the patients with PAH, like pulmonary blood volume, blood flow and perfusion heterogeneity, can be determined.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a rare, life-threatening disease. It is characterized by the elevation of pulmonary arterial pressure and pulmonary vascular resistance. A remodeling of small pulmonary vessels characterized by the proliferation of the adventitia, the hypertrophy of the media and fibrosis of the intima can be observed on the microscopic level.

Non-invasive techniques for hemodynamic assessment and identification of early pulmonary vascular remodeling and pulmonary hypertension have a marked practical advantage as compared to invasive right heart catheterization, however, their accuracy and reliability is not well established.

In the present study the investigators examine patients who are scheduled for a thorax CT with an additional dynamic contrast-enhanced DE-CT protocol and derive established parameters for the diagnosis of PAH as well as novel parameters from the CT scans. These are compared to results from the right-heart catheterization and other investigations routinely carried out on these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with right heart catheterization data

Exclusion Criteria:

* patients with decreased renal function
* patients who received CT in the previous six months
* intolerance of contrast material
* other standard CT contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary blood flow and volume determined by dual energy computed tomography | measurements with right heart catheterisation within 1 month
  validation of pulmonary blood flow and volume of pulmonary hypertension patients

SECONDARY OUTCOMES:
Comparison of dual energy computed tomography derived data with clinical findings of pulmonary hypertension patients | measurements with right heart catheterisation within 1 month
  comparison of different state or type of pulmonary hypertension
Lung perfusion heterogeneity determined by dual energy computed tomography | measurements with right heart catheterisation within 1 month
  quantification of regional perfusion differences in pulmonary hypertension patients

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Division of Pulmonology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No